CLINICAL TRIAL: NCT01254266
Title: Morbid Obesity in Children and Adolescents : Does Inpatient Treatment in a Psychosomatic Unit Increases the Chance for a Long-term Weight Maintenance?
Brief Title: The Efficacy of an Inpatient Program for Long-term Weight Maintenance in Children and Adolescents With Morbid Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Silvana Fennig, M.D., Rabin Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5833
Record Dates: First submitted 2010-11-09; First posted 2010-12-06 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2010-05

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; adolescents; inpatient treatment
MeSH Terms: conditions — Obesity, Morbid | interventions — Length of Stay; Hospitalization; Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conservative treatment (Experimental): conservative weight reduction treatment in an inpatient unit.
  Interventions: Behavioral: inpatient hospitalization and follow up; Behavioral: inpatient treatment and follow up
- bariatric surgery (Experimental): inpatient program as a pre- and post- operational 'envelope' for bariatric surgeries.
  Interventions: Procedure: bariatric surgery; Behavioral: inpatient treatment with follow up

INTERVENTIONS:
Behavioral: inpatient hospitalization and follow up — An inpatient program and a 1-year weekly follow up that include multi-disciplinary interventions for weight reduction and maintenance.
  Arms: conservative treatment
Behavioral: inpatient treatment and follow up — one month inpatient treatment followed by a year-long follow up on the inpatient unit.
  Arms: conservative treatment
Procedure: bariatric surgery — bariatric surgery.
  Arms: bariatric surgery
Behavioral: inpatient treatment with follow up — 1 month inpatient treatment followed by a year-long follow up on the inpatient unit.
  Arms: bariatric surgery

SUMMARY:
The major problem in the treatment of morbidly obese children is the long term maintenance of the reduced weight. Maintenance-focused interventions have not been studied enough in adolescents with morbid obesity, neither in regard to conservative methods of weight reduction, nor in regard to bariatric surgeries.

This study will investigate the effectiveness of an integrative, multi-disciplinary inpatient program for promoting long-term weight maintenance in children with morbid obesity. The program will be studied in two perspectives: as a conservative treatment, as well as an 'envelope' for bariatric surgeries including a pre-operational preparation phase and a post-operational follow-up.

The investigators hypothesize that program participants will maintain weight significantly better than the proportion known in the literature.

DETAILED DESCRIPTION:
Background: The major problem in the treatment of morbidly obese children and adolescents is not weight reduction itself, but the long term maintenance of the reduced weight. Treatment of morbid obesity has a dual goal: Immediate relief for the obesity-related physical symptoms (by moderate weight reduction), and prevention of relapse by encouraging weight maintenance. Without maintenance-focused interventions, morbidly obese children are prone for repeated weight gains that can induce further complications and undermine therapeutic efforts. Maintenance-focused interventions have not been studied enough in adolescents with morbid obesity. An alternative solution for the conservative approach described above is based on bariatric surgeries. These are currently limited in adolescents due to insufficient evidence regarding pre- and post-operational interventions for long term weight maintenance.

Goals: The study is designed to investigate the effect of an integrative, multi-disciplinary program for children and adolescents with morbid obesity. The program includes interventions for moderate weight reduction and for long term weight maintenance. The program is based on a year-long treatment continuum. The different phases of this continuum include a short hospitalization, intensive day treatment program, and weekly follow up. The program is also based on intensive work with parents, with emphasis on familial change of life habits. The program will be studied in two perspectives: as a conservative treatment, as well as an 'envelope' for bariatric surgeries including a pre-operational preparation phase and a post-operational follow-up.

Hypothesis: The proportion of program participants who will decrease their weight and maintain it for at least one year will be significantly higher than the proportion known in the literature. This finding is expected among participants in the 'conservative' program as well as among participants who will undergo bariatric surgeries.

Method: the study will take place in a child and adolescent psychiatric unit located in a general children hospital, in cooperation with pediatric and endocrinology units. Participants will undergo short hospitalization focused on acute relief of obesity related complications and as a pre-operational preparation for those participants who are designated for surgery. All participants, whether designed for operation or not, will continue participation in a year long day program focused on weight maintenance and acquisition of healthy life habits. Study design will include 4 assessments of psychical and psychological measures: pre-hospitalization screening, admission, 4-month follow up, 1-year follow up. At those assessment points, both children and parents will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. BMI > 40, with a physical complication known to improve by weight reduction or BMI > 95% for age and weight with a serious obesity-related physical complication that without intervention would require acute invasive procedure.
2. Previous failures in obtaining weight reduction in the framework of intensive, outpatient programs.
3. Voluntary participation by the child and his or her family and high motivation for change as assessed in a pre-hospitalization assessment.

Exclusion Criteria:

1. Failure of parents in applying changes required by the program (e.g., missing parent guidance appointments).
2. Lack of cooperation with the program (e.g., non-compliance with dietary regime, failure in maintaining food diaries).
3. Failure to obtain weight reduction in two consecutive weeks, without a clear physical or medical cause.

   -

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Weight | 1 year from hospitalization
  The subject's weight will be measured.

SECONDARY OUTCOMES:
Weight | Pre-hospitalization screening, admission, and 4-month follow-up.
  Subject's weight will be measured.
Clinical condition, as measured in an adapted version of the Morgan-Russel scale. | pre-hospitalization screening, admission, 4-month follow-up, and 1-year follow-up.
  The clinical features of morbid obesity and symptoms of other eating disorders are assessed using a semi-structured clinical interview.
Endocrinological and physical condition | admission, 4-month follow-up, and 1-year follow-up.
  Blood Tests: SMA (including fasting glucose, and lipid profile), blood cell count, HBA1c, TSH, FT4, Folic Acid, Fasting Insulin, B12, Forum. Urine Cortisol. In Acanthosis Nigricans, Hyperlipidemia, or high Blood Pressure, an OGTT test will be performed. In abnormal hepatic enzymes, an abdominal ultrasound will be performed. In menstrual abnormalities additional blood tests will be performed:LH, FSH,Andostrindione, Testosterone,17 OHP, DEHAS. Physical Examination and Diagnostic Tests: BIA (Bioelectrical Bioimpedance Analysis),skinfold thickness measurement, Blood Pressure , EKG.
Depression as measured by the Beck Depression Inventory (BDI). | pre-hospitalization screening, admission, 4-month follow-up, and 1-year follow-up.
  The BDI is a valid and reliable measure of depression.
Psychological features association with eating disorders measured by Eating Disorders Inventory - 2(EDI-2) | Pre-hospitalization assessment, admission, 4-month follow-up and 1-year follow-up.
  The EDI-2 is a valid and reliable measure of psychological features of eating disorders.
Symptoms of morbid obesity and eating disorders as measured by the Eating Disorders Examination, questionnaire version (EDE-Q). | Admission, 4-month follow-up, and 1-year follow-up.
  The EDE-Q will be administered as a self-report questionnaire. It is a valid and reliable measure of symptoms of eating disorders and obesity.
Self-efficacy, as measured by the self-efficacy questionnaire. | pre-hospitalization screening, admission, 4-month follow-up, and 1-year follow-up.
  Subject's self-efficacy to control behaviors and feelings realted to obesity and management of weight. The self-efficacy questionnaire was written for this study.
Motivation for treatment, as measured by the Treatment Motivation Scale (TMQ). | pre-hospitalization screening, admission, 4-month follow-up, and 1-year follow-up.
  The TMQ is a valid and reliable measure to assess motivation for treatment.
Life Habits. | pre-hospitalization screening, and 4-month follow-up.
  Life habits will be assessed using a semi-structured interview designed easpecially for the purpose of the current study. The interview includes questions about eating behaviors, family life style, living arrangements, patterns of food consumption and availability etc.
Structured Clinical Interview for Axis I DSM-IV Disorders (SCID). | pre-hospitalization screening.
  The SCID is a semi-structured interview designed to assess and diagnose the presence of Axis I disorders.
Clinical Demographic Questionnaire | pre-hospitalization screening.
  This questionnaire assess demographic information as well as information regarding weight history, development of diatery regime, as well as previous treatment and/or hospitalization.
Parent's Self-efficacy, as measured by the parent's self-efficacy questionnaire. | pre-hospitalization screening, admission, 4-month follow-up, and 1-year follow-up.
  Parent's self-efficacy to help his or her child to control behaviors and feelings realted to obesity and management of weight. The parent's self-efficacy questionnaire was written for this study.
Child's motivation for treatment, from the perspective of the parent. | pre-hospitalization screening, admission, 4-month follow-up, and 1-year follow-up.
  The parent's view on the child's motivation for treatment. This variable will be measured using an adapted veriou of the Treatment Motivation Scale (TMQ).
Parent's depression as measured by the Beck Depression Inventory (BDI). | pre-hospitalization screening, admission, 4-month follow-up, and 1-year follow-up.
  The BDI is a valid and reliable measure of depression.
Parent's Clinical Demographic Questionnaire | pre-hospitalization screening.
  This questionnaire assess demographic information as well as information regarding child's weight history, development of diatery regime, as well as previous treatment and/or hospitalization.
Child's clinical condition, from the perspective of the parent. | pre-hospitalization screening, admission, 4-month follow-up, and 1-year follow-up.
  The clinical features of morbid obesity and symptoms of other eating disorders are assessed using a semi-structured clinical interview based on and adaptation of the well-establised Morgan-Russel Scale.
Child's life habits, from the perspective of the parent. | pre-hospitalization screening, and 1-year follow-up.
  Life habits will be assessed using a semi-structured interview designed easpecially for the purpose of the current study. The interview includes questions about eating behaviors, family life style, living arrangements, patterns of food consumption and availability etc.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Fennig, M.D., Principal Investigator — Rabin Medical Canter; Tamar Tahar, R.N., Study Director — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel